CLINICAL TRIAL: NCT05190510
Title: Assessment of Vulnerability to Carotid Stenosis by MultiModal Imaging and Cellular and Molecular Biology Analysis Pilot Study
Brief Title: Assessment of Vulnerability to Carotid Stenosis by MultiModal Imaging and Cellular and Molecular Biology Analysis
Acronym: EVA3M
Status: Terminated | Type: Observational
Why Stopped: The carotid plaque is too small to quantify activity with the standard protocol used, despite a rigorous protocol and methodology.
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: STEINMETZ 2021
Record Dates: First submitted 2021-10-11; First posted 2022-01-13 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Internal Carotid Artery; Atheromatous Stenosis
MeSH Terms: interventions — Data Collection; Cell Count; Gene Expression Profiling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — collection of the carotid plaque (surgical specimen)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with atheromatous stenosis of the internal carotid artery
  Interventions: Other: Data collection; Procedure: collection of the carotid plaque (surgical specimen); Other: anatomopathological, histological, cellular and molecular biology examinations (metabolomics and transcriptomics) on surgical specimens

INTERVENTIONS:
Other: Data collection — Collection of data from preoperative imaging examinations (routine examination prescribed before the operation)
Procedure: collection of the carotid plaque (surgical specimen) — collection of the carotid plaque
Other: anatomopathological, histological, cellular and molecular biology examinations (metabolomics and transcriptomics) on surgical specimens — anatomopathological, histological, cellular and molecular biology examinations (metabolomics and transcriptomics) on surgical specimens

SUMMARY:
Cerebrovascular accidents (CVA) are the second leading cause of death in France, and the most frequent cause of acquired physical and mental disability. Up to 90% of strokes are ischemic, among which about 15% are due to the presence of stenosis of the carotid sinus, at the base of the extracranial internal carotid artery.

For many years, only the degree of stenosis was used to assess the risk of stroke, based on the results of original studies from the 1990s. However, the significant improvement in medical treatments since then has significantly reduced the risk of stroke, and the benefits of carotid intervention are becoming increasingly debatable.

Since the publication of the latest recommendations, the degree of stenosis alone is no longer sufficient to propose an intervention, since most of them will never lead to a neurological event. In addition to stenosis greater than 60%, for the first time, other criteria must be sought to decide on treatment. For example, so-called carotid plaque "vulnerability" criteria, defining patients "at high risk of stroke," should be sought.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic or asymptomatic atheromatous stenosis of the internal carotid artery, of a degree ≥ 50%, for which an operative indication is retained
* Scheduled surgery

Exclusion Criteria:

Samples collected from patients :

* who did not have a preoperative CT angiogram of the supra-aortic trunks
* with contraindication to MRI
* with contraindication to PET scan
* with a history of cervical radiotherapy
* with uncontrolled diabetes
* with a previous homolateral carotid endarterectomy
* who has already undergone angioplasty-stenting of the homolateral carotid artery
* with a neoplasia considered active / not cured
* Surgical procedure performed in emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Scheduled surgery
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
rate of 18FDG tracer uptake in carotid stenosis | At baseline
Degree of instability of the plate | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France